CLINICAL TRIAL: NCT05455931
Title: Prospective Research Based Observational Study of Poteligeo® Experience in the Real World in Adult Patients With Mycosis Fungoides and Sézary Syndrome
Brief Title: Real World Observational Study of Poteligeo in Adult Patients With MF and SS (PROSPER)
Acronym: PROSPER
Status: Active, not recruiting | Type: Observational
Sponsor: Kyowa Kirin Pharmaceutical Development Ltd (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Other Study IDs: 2022-05-WW-POT
Record Dates: First submitted 2022-07-04; First posted 2022-07-13 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Mycosis Fungoides and Sézary Syndrome
MeSH Terms: conditions — Mycosis Fungoides; Sezary Syndrome | interventions — mogamulizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with MF/SS: Adult patients with diagnosed MF/SS receiving Poteligeo treatment.
  Interventions: Drug: Poteligeo

INTERVENTIONS:
Drug: Poteligeo — Poteligeo treatment will be used as prescribed by the Investigator in accordance with the terms of the reimbursed indication within the relevant country. The assignment of the patient to a particular therapeutic strategy falls within current practice and the prescription of Poteligeo is clearly separated from the decision to include the patient in the study.
  Other Names: Mogamulizumab

SUMMARY:
This is a prospective, observational, non-interventional, international, multi-center, mixed methods study that will involve the integration of quantitative and qualitative data in patients with MF/SS treated with Poteligeo.

DETAILED DESCRIPTION:
The PROSPER study aims to collect information about the experiences of patients with MF/SS receiving Poteligeo and of their caregivers in real-world clinical practice. The objective of this study is to generate patient-level data to provide insights into real world clinical practice and an understanding of treatment decisions, as well as to collect patient reported outcomes (PRO) data, enriched with qualitative data on disease and treatment experience and burden, to demonstrate the full impact of treatment and the relevant patient experience in real-world clinical practice. The study will be conducted 6 countries, including North America, United Arab Emirates and countries in Europe, at 19 sites known to treat and follow-up patients with MF/SS. Patients will be followed for up to 50 weeks from study enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged ≥18 years
2. Confirmed diagnosis of MF/SS
3. Disease staging at enrollment has been completed
4. About to commence primary treatment with Poteligeo® as per reimbursed indication
5. Patient is willing and able to complete the symptom diary and PROs.
6. Patient is willing and able to provide written informed consent to participate in the study in a manner approved by Institutional Review Board(IRB)/ Independent Ethics Committee (IEC) and local regulations

Exclusion Criteria:

1. Patient unable to participate in all aspects of the study and/or does not agree to the collection of data from medical records
2. Patient currently participating in an interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 80 patients with a confirmed diagnosis of MF/SS and about to commence primary treatment with Poteligeo as per reimbursed indication will be recruited from approximately 19 sites across North America, United Arab Emirates and Europe.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2025-08-07 (Estimated); Study Completion 2025-08-07 (Estimated)

PRIMARY OUTCOMES:
To describe the patient-reported change in key signs and symptoms of disease following initiation of treatment with Poteligeo. | Weekly for first 16 weeks, then every 4 weeks until Week 48, at treatment discontinuation and 8 and 16 weeks after treatment discontinuation.
  Patients will complete a symptom diary at regular intervals throughout the study to record symptoms including skin pain, skin itch, skin flaking, skin redness, difficulty regulating body temperature and sleep problems.
To describe the patient-reported change in fatigue following initiation of treatment with Poteligeo. | Every 12 weeks from first dose visit to treatment discontinuation and then 8 and 16 weeks after treatment discontinuation.
  Patients will complete PRO questionnaire BFI to assess changes in fatigue
To describe the patient-reported change in health-related QoL following initiation of treatment with Poteligeo. | Every 12 weeks from first dose visit to treatment discontinuation and then 8 and 16 weeks after treatment discontinuation.
  Patients will complete PRO questionnaire CTCL-QoL at regular time points throughout the study to assess any changes in quality of life.
To assess change in the HRQoL of the patient's main caregiver | First dose visit, at week 12 after the first Poteligeo® administration, and within 4 weeks of treatment discontinuation.
  The patient's main caregiver will be invited to complete the CareGiver Oncology Quality of Life questionnaire (CarGOQoL)

CONTACTS AND LOCATIONS:
Overall Officials: Kyowa Kirin Medical Affairs Division, Study Director — Kyowa Kirin Medical Affairs Division
Locations (19):
- United States (5):
  - The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Colombia University Medical Center, New York, New York
  - Inova Dwight and Martha Schar Cancer Institute, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Italy (6):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Do Ancona, Ancona
  - IRCCS A.O.U. Policlinico S. Orsola - Malpighi, Bologna
  - Azienda Ospedaliero- Universitaria Careggi, Florence
  - Ematologia Policlinico di Milano, Milan
  - IFO-San Gallicano IRCCS, Rome
  - Universita Cattolica del Sacro Cuore - Policlinico Universitario Agostino Gemelli, Rome
- Leids Universitair Medisch Centrum (LUMC), Leiden, Netherlands
- Spain (2):
  - Hospital Del Mar, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
- Sheikh Shakhbout Medical City, Abu Dhabi, United Arab Emirates
- United Kingdom (4):
  - Clatterbridge Hospital - Wirral University Teaching Hospital Nhs Foundation Trust, Bebington
  - University Hospital Birmingham, Birmingham
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust - Nottingham City Hospital, Nottingham